CLINICAL TRIAL: NCT04572802
Title: Study on the Changes of Serum Orphanin FQ in Patients With Diabetes Mellitus and Coronary Heart Disease in Different Courses
Brief Title: Changes of Serum Orphanin FQ in Patients With Coronary Heart Disease in Different Courses of Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, principal investigation, Second Hospital of Shanxi Medical University
Other Study IDs: hanyi20200802
Record Dates: First submitted 2020-09-29; First posted 2020-10-01 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Type2 Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum orphanin FQ,Glycosylated hemoglobin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- control group: Coronary heart disease population: after coronary angiography, Gensini score was used to evaluate the severity of coronary artery occlusion, and then compared with the population of type 2 diabetes complicated with coronary heart disease
  Interventions: Procedure: Coronary angiography
- experimental group (course of disease <5 years): Type 2 diabetes complicated with coronary heart disease (course of disease 5-10 years).Retrospective examination of patients' data, recording patients' laboratory tests and drug use, taking blood to measure orphanin, and evaluating the severity of coronary artery occlusion with Gensini score.
  Interventions: Procedure: Coronary angiography
- experimental group(course of disease 5-10 years): Type 2 diabetes complicated with coronary heart disease (course of disease 5-10 years).
  Interventions: Procedure: Coronary angiography
- experimental group(course of disease10-20 years): Type 2 diabetes complicated with coronary heart disease (course of disease 10 -20years).Finally, the data were obtained to evaluate the relationship between the course of diabetes and the severity of coronary heart disease, as well as the relationship between the course of diabetes and OFQ in patients' blood.
  Interventions: Procedure: Coronary angiography

INTERVENTIONS:
Procedure: Coronary angiography — Coronary angiography was performed in patients with coronary heart disease complicated with type 2 diabetes mellitus

SUMMARY:
To explore the severity of diabetic patients with coronary heart disease and the change of serum orphanin FQ content in different diabetic courses

DETAILED DESCRIPTION:
Methods: A retrospective case-control study was conducted. The control group was a patient who underwent coronary angiography at the same time and was definitely diagnosed as coronary heart disease but not diabetes. The study group was coronary heart disease complicated with diabetes, which was divided into group A (≤5 years), group B (5-10 years) and group C (10-20 years) according to the course of diabetes. (1) Review the electronic medical records and record the general information of the selected patients: age, sex, history of hypertension, history of myocardial infarction, family history of coronary heart disease, smoking history, chronic kidney disease; ② laboratory findings: HbA1C (glycosylated hemoglobin), SBP (systolic blood pressure), DBP (diastolic blood pressure), total cholesterol, HDL, LDL, triglyceride, BMI, creatinine and glomerular passing rate (EGFR); ③ Drug use: oral hypoglycemic agents, insulin, aspirin, statins, hypertension drugs, ACEI or ARB, β-blockers, CCB and diuretics. (ii) Taking coronary angiography as the gold standard, the grading index of severity of coronary heart disease was made, and the severity of coronary heart disease was evaluated by Gensini score.

ELIGIBILITY:
Inclusion Criteria:

* The main discharge diagnosis is T2DM；;
* Age > 18 years old;
* No acute complications of diabetes;
* The previous diagnosis was coronary heart disease

Exclusion Criteria:

* T1DM patients;
* EGFR < 60 ml/min/1.73 m or proteinuria (or both);
* Patients with history of acute cardiovascular events;
* Familial hypercholesterolemia or other hereditary lipid metabolism diseases;
* anti-HIV patients;
* Patients with serious mental health problems;
* Patients receiving drugs that can lead to dyslipidemia, such as antipsychotics, corticosteroids, or immunosuppressants;
* Patients with systemic inflammatory diseases, such as systemic lupus erythematosus; Pet-name ruby is quitting smoking and severe obesity (BMI>40).

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes complicated with coronary heart disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Gensini score | 1 week
  Gensini score was used to evaluate the severity of coronary artery occlusion, and then compared with the population of type 2 diabetes complicated with coronary heart disease

CONTACTS AND LOCATIONS:
Overall Officials: zheng guo, doctor, Principal Investigator — Second Hospital of Shanxi Medical University
Locations (1):
- Second of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
All IPD that underlie results in a publication